CLINICAL TRIAL: NCT00527579
Title: PET Imaging of Peripheral Benzodiazepine Receptors in Patients With Neurocysticercosis Using [F-18]FBR
Brief Title: PET Imaging of Peripheral Benzodiazepine Receptors in Patients With Neurocysticercosis Using [F-18]FB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 070209; 07-M-0209
Record Dates: First submitted 2007-09-08; First posted 2007-09-11 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2013-11-26

CONDITIONS: Neurocysticercosis; Healthy
Keywords: Epilepsy; Taenia Solium; Microglia; Neuroinflammation; Compartment Model; Neurocysticercosis; Healthy Volunteer; HV
MeSH Terms: conditions — Neurocysticercosis; Epilepsy; Taeniasis; Neuroinflammatory Diseases

INTERVENTIONS:
Drug: [F-18]FBR

SUMMARY:
The purpose of this protocol is to measure peripheral benzodiazepine receptors in the brain using positron emission tomography (PET) and compare the imaging results between patients and healthy people.

DETAILED DESCRIPTION:
Objective

In endemic regions neurocysticercosis is the most common cause of adult acquired epilepsy and thus an important public health problem. The disease is caused by infection with the larval form of the tapeworm, Taenia solium. Although neurocysticercosis is common only in many developing regions, an increased number of patients are diagnosed in developed countries mostly due to immigration of infected individuals.

The peripheral benzodiazepine receptor (PBR) can be a clinically useful marker to detect neuroinflammation because activated microglia in inflammatory areas expresses high levels of PBR. PBR has been imaged with positron emission tomography (PET) using [(11) C]1-(2-chlorophenyl-N-methylpropyl)-3-isoquinoline carboxamide (PK11195), which provides low levels of specific signal. Recently we developed a new ligand, N-fluroacetyl-N-(2,5-dimethoxybenzyl)-2-phenoxyaniline ([(18)F]FBR), which showed much greater specific signals than [(11) C]PK11195 in non-human primates.

The major objective of this protocol is to assess the utility of [(18) F]FBR PET to detect neuroinflammation in patients with neurocysticercosis.

A secondary objective is to study whether some healthy subjects do not show binding of [(18)F]FBR by performing whole body imaging using [18F]FBR and binding assays using blood cells. In other protocols using a PET ligand with similar structure, [(11)C]PBR28, approximately 8% of subjects (9/~ 118 ) did not show binding. In protocols 07-N-0035 and 08-M-0158, we compared binding of [11C]PBR28 and [(11)C]PK 11195 in approximately ten healthy subjects including five who did not show binding of [(11)C]PBR28 in prior whole body imaging. We found differences in organs with regard to sensitivity to the phenomenon of non-binding. In the non-binders, PBR28 showed no binding in all five organs with high PBR density. However, PK 11195 showed significantly reduced binding in only two organs with PBR. We now wish to determine whether PBR06 is more similar to PBR28 or to PK 11195 in terms of the non-binding phenomenon. In the current protocol, in addition to whole body imaging using [(18)F]FBR, we will do in vitro binding assays using blood cells as another tissue to examine the effect of non-binding.

Study population

For [(18)F]FBR brain scans, ten patients will be recruited and clinically followed under protocol 85-I-0127, Treatment of Cysticercosis including Neurocysticercosis with Praziquantel or Albendazole (PI: Theodore E. Nash, MD, NIAID). Fifteen healthy subjects will be recruited.

For whole body scan using [(18)F]FBR, additional 30 healthy subjects will be recruited. Therefore, total accrual numbers are 10 patients with neurocysticercosis and 45 healthy subjects (15 for brain [(18)F]FBR and 30 for whole body [(18)F]FBR scans.

Design

Ten patients with neurocysticercosis and 15 age-matched healthy subjects will have brain PET scans. In addition, we will also perform a whole body PET scan on 30 healthy subjects to study the radiation-absorbed doses and study whether some healthy subjects do not show binding of [(18)F]FBR. Patients will have up to three [(18)F]FBR PET scans during the follow-up and the treatment under 85-I-0127, typically a few weeks apart.

Outcome measures

<TAB>

In brain PET scans, [(18)F]FBR binding will be compared with clinical symptoms and MRI findings. In addition, the binding will be compared between patients and age-matched control subjects. We have calculated radiation absorbed doses in approximately seven healthy subjects who showed normal distribution (i.e., binders) of activity in organs. If we found subjects who appear to have no binding to [(18)F]FBR, we will calculate radiation-absorbed doses of the non-binders.

ELIGIBILITY:
* INCLUSION CRITERIA:

COMMON TO PATIENTS WITH NEUROCYSTICERCOSIS AND HEALTHY SUBJECTS:

Ages between 18 and 65, inclusive.

<TAB>

In addition, patients must meet the inclusion criteria of protocol 85-I-0127.

Control subjects are healthy based on history, physical exams, ECG, and lab tests.

EXCLUSION CRITERIA:

COMMON TO ALL SUBJECTS:

Current psychiatric illness, substance abuse or severe systemic disease based on history and physical exam.

ECG with clinically significant abnormalities. Any existing physical exam and ECG within one year will be reviewed and if none already exists in the chart, these will be obtained and reviewed.

Prior participation in other research protocols or clinical care in the last year such that radiation exposure would exceed the annual guideline of RSC.

Pregnancy or breast feeding.

Claustrophobia.

Positive HIV test.

Cannot lie on back for a few hours for the PET scans.

ADDITIONAL EXCLUSION CRITERIA TO BRAIN SCANS:

Presence of ferromagnetic metal in the body or heart pacemaker.

[(18)F]FBR did not show binding in a whole body PET [(18)F]FBR scan in the past.

ADDITIONAL EXCLUSION CRITERIA FOR PATIENTS:

Medically unstable.

Seizures are not well controlled with medications.

A history of brain disease other than neurocysticercosis.

Laboratory tests with clinically significant abnormalities unrelated to neurocysticercosis or its treatment.

ADDITIONAL EXCLUSION CRITERIA FOR HEALTHY SUBJECTS:

Laboratory tests with clinically significant abnormalities.

A history of brain disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-09-04; Primary Completion 2013-11-26 (Actual); Study Completion 2013-11-26 (Actual)

PRIMARY OUTCOMES:
Binding of [F-18]FBR at peripheral benzodiazepine receptor. | 3 years

SECONDARY OUTCOMES:
MRI | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Fujita, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Anholt RR, De Souza EB, Oster-Granite ML, Snyder SH. Peripheral-type benzodiazepine receptors: autoradiographic localization in whole-body sections of neonatal rats. J Pharmacol Exp Ther. 1985 May;233(2):517-26. PMID 2987488
- [Background] Anholt RR, Murphy KM, Mack GE, Snyder SH. Peripheral-type benzodiazepine receptors in the central nervous system: localization to olfactory nerves. J Neurosci. 1984 Feb;4(2):593-603. doi: 10.1523/JNEUROSCI.04-02-00593.1984. PMID 6321699
- [Background] Anholt RR, Pedersen PL, De Souza EB, Snyder SH. The peripheral-type benzodiazepine receptor. Localization to the mitochondrial outer membrane. J Biol Chem. 1986 Jan 15;261(2):576-83. PMID 3001071